CLINICAL TRIAL: NCT00100854
Title: A Randomized, Open-Label Phase II Clinical Trial of Combination Erlotinib (Tarceva®) and Fulvestrant (Faslodex®) Versus Erlotinib (Tarceva®) Alone in Advanced Non-Small Cell Lung Cancer Patients
Brief Title: Erlotinib With or Without Fulvestrant in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Oncology Research International (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000407580; P50CA090388 (NIH); P30CA016042 (NIH); UCLA-0407058-01
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive oral erlotinib hydrochloride once daily on days 1-28. Courses repeat every 28 days.
  Interventions: Drug: erlotinib hydrochloride
- Arm II (Experimental): Patients receive erlotinib hydrochloride as in arm I and fulvestrant intramuscularly on days 1, 15, and 29, and then every 28 days thereafter.
  Interventions: Drug: erlotinib hydrochloride; Drug: fulvestrant

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
Drug: fulvestrant — Given intramuscularly
  Arms: Arm II

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of non-small cell lung cancer cells. Hormone therapy using fulvestrant may fight non-small cell lung cancer by lowering the amount of estrogen the body makes. Giving erlotinib together with fulvestrant may kill more tumor cells. It is not yet known whether giving erlotinib together with fulvestrant is more effective than erlotinib alone in treating non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying giving erlotinib together with fulvestrant to see how well it works compared to erlotinib alone in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare objective tumor response in patients stage IIIB or IV non-small cell lung cancer treated with erlotinib hydrochloride with vs without fulvestrant.

Secondary

* Correlate response rate with ER and EGF receptor expression in patients treated with these regimens.
* Correlate measurement of ER-α, ER-β, EGF/HER-1 receptor and HER-2/neu receptor with clinical response in patients treated with these regimens.
* Correlate erlotinib hydrochloride resistance with ER and HER receptor expression in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to performance status, gender, and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral erlotinib hydrochloride once daily on days 1-28. Courses repeat every 28 days.
* Arm II: Patients receive erlotinib hydrochloride as in arm I and fulvestrant intramuscularly on days 1, 15, and 29, and then every 28 days thereafter.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 30 days and then every 2 months until disease progression.

PROJECTED ACCRUAL: A total of 102 patients (34 in arm I and 68 in arm II) will be accrued for this study.

ELIGIBILITY:
Inclusion criteria:

* adults over the age of 18 capable of giving informed consent.
* Histologically confirmed non-small cell lung cancer
* Stage IIIB or IV NSCLC
* Tumor tissue block available.
* ECOG performance status of 0, 1 or 2.
* Measurable disease by RECIST criteria defined as ≥ 1 target lesion that has not been irradiated. New lesions that have developed in a previously irradiated field may be used as sites of measurable disease provided all other criteria are met.
* Meets 1 of the following criteria:
* Progressive disease after ≥ 1 prior standard chemotherapy regimen
* Refused chemotherapy
* Unable to receive standard chemotherapy
* women of childbearing age must have negative pregnancy test by urine or serum prior to initiation of treatment. men and women of childbearing potential must consent to using adequate contraception throughout treatment and for 3 months following surgery.

Exclusion criteria:

* Renal insufficiency (serum creatinine >2mg/dl)
* Liver insufficiency (serum total bilirubin >1.5X ULN, or serum transaminases > 2.5X the ULN or %X ULN if hepatic metastases).
* hematologic abnormality platelets< 100,000 ANC <1,500/mm3
* THerapeutic anticoagulation will be allowed, but patients receiving fulvestrant while on therapeutic anticoagulation will have the fulvestrant dose divided into twice as many syringes to minimize the volume of intramuscular injection in these patients. In patients receiving low molecular weight heparin or fondaparinux, these medications should be held for 12 hours before and after fulvestrant injection if possible.
* Active CNS metastases.
* New York Heart Association class III or IV cardiac disease
* myocardial infarction within the past 12 months
* symptomatic ventricular arrhythmia
* symptomatic conduction abnormality
* evidence of clinically active interstitial lung disease
* Patients with asymptomatic chronic stable radiographic changes are eligible
* pregnant or nursing or inadequate contraception
* hypersensitivity to erlotinib hydrochloride or fulvestrant or to any of their excipients
* comorbid disease or medical condition that would preclude study treatment or compliance
* malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* chemotherapy or non-cytotoxic investigational agents within 4 weeks of initiating treatment.
* major surgery within 4 weeks of initiating therapy. Minor surgery within 7 days of initiating therapy.
* anticancer antiestrogen therapy. Concurrent stable-dose steroids allowed
* concomitant radiation therapy to the lungs. Radiation therapy to non-target lesions will be allowed as long as it is completed 1 week prior to initiation of treatment.
* prior anticancer epidermal growth factor receptor inhibitors
* concurrent CYP3A4 inducers, including any of the following:
* Phenytoin
* Carbamazepine
* Rifampin
* Barbiturates
* Hypericum perforatum (St. John's wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2004-10-28 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Objective tumor response | 30 days

SECONDARY OUTCOMES:
Correlation of response rate with receptor expression | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Edward Garon, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States